CLINICAL TRIAL: NCT01910324
Title: Facilitating Adolescent Offenders' Reintegration From Juvenile Detention to Community Life (DTC)
Brief Title: Juvenile Detention to Community Life
Acronym: DTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Howard Liddle, Professor, University of Miami
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 20043161
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Substance Use; Delinquency; Risk for HIV Infection
Keywords: Juvenile Offenders; HIV/STD Prevention; Adolescent Substance Abuse; Multidimensional Family Therapy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multidimensional Family Therapy Cross-Systems (Experimental): In Stage 1 (in detention) Multidimensional Family Therapy Cross-Systems (MDFT-CS) consists of two major components: standard initial/engagement work with parents in the home and with adolescents in detention, plus a state-of-the-art HIV education prevention module. In Stage 2, MDFT-CS includes the standard MDFT components: 1) interventions with the adolescent, 2) interventions with the parent, 3) interventions to improve the parent-adolescent relationship, 4) interventions with other family members, and 5) interventions with external systems.
  Interventions: Behavioral: Multidimensional Family Therapy Cross-Systems
- Enhanced Services as Usual (Other): In Stage 1 (in detention) ESAU includes two major components: standard drug treatment services delivered by detention staff, and state-of-the-art HIV education prevention intervention. In Stage 2, community drug treatment providers deliver high quality drug treatment on an outpatient basis.
  Interventions: Behavioral: Enhanced Services as Usual

INTERVENTIONS:
Behavioral: Multidimensional Family Therapy Cross-Systems — Standard initial/engagement work in the home and detention, plus a state-of-the-art HIV education prevention module as well as standard MDFT which assesses and intervenes in five domains: 1) Interventions with the adolescent, 2) interventions with the parent, 3) interventions to improve the parent-adolescent relationship, 4) interventions with other family members, and 5) interventions with external systems.
  Other Names: MDFT-CS
  Arms: Multidimensional Family Therapy Cross-Systems
Behavioral: Enhanced Services as Usual — Standard drug treatment services in detention and state-of-the-art HIV education prevention intervention, as well as outpatient drug treatment provided by community drug treatment providers
  Other Names: ESAU
  Arms: Enhanced Services as Usual

SUMMARY:
The fundamental objective of the proposed study is to develop and test an innovative two-stage, cross-systems family-based intervention for substance abusing juvenile offenders. The first stage of the experimental treatment is provided for youths in juvenile detention settings. Stage two of the intervention occurs after the offender is released to the community. Participants are randomized to one of two study conditions: the cross-systems family-based intervention (Multidimensional Family Therapy-Cross Systems (MDFT-CS), or 2) Enhanced Services as Usual (ESAU). Both conditions incorporate HIV prevention in detention and we will also examine the effects of a family-based HIV/STD prevention module beyond the impact of a standard HIV/STD education intervention delivered in detention by including ongoing HIV/STD intervention in MDFT-CS following release from detention. There are five aims of the proposed study. These aims relate to: 1) Intervention development and implementation; 2) Clinical effectiveness; 3) Impact of HIV/AIDS/STD prevention; 4) Comparative benefit-costs; and 5) Systems-level impact

DETAILED DESCRIPTION:
This study will employ a fully randomized (2 conditions) by 9 assessment points (baseline, discharge from detention, and 3, 6, 9, 18, 24, 36 and 42 months following detention discharge), repeated measures intent-to-treat design with multiple dependent variables. 154 males and females (85 participants from Miami Dade Regional Juvenile Detention Center and 85 from Pinellas Juvenile Detention Center) who meet the study eligibility criteria will be randomized to one of the two treatment conditions.

The study will also include a 6-month pilot phase. During this phase, the MDFT detention intervention and cross-systems collaboration protocols will be developed; the existing treatment manual will be revised; the MDFT-CS with family-based HIV prevention module and standard HIV education intervention will be developed; family therapists will be trained in the MDFT intervention (including HIV/STD module); the MDFT-CS intervention will be piloted; the assessment battery will be piloted; the protocols, manual, and training package will be revised and finalized; research staff will be trained on all procedures and protocols; and data management procedures will be developed.

During Stage 1, adolescents in all intervention conditions will receive standard detention services, which include education and health care. In addition, youth assigned to the ESAU condition will receive the standard mental health and substance abuse services offered in the detention (mainly psychoeducational in nature). Youth assigned to the MDFT-CS intervention will not receive standard mental health/substance abuse services provided by the detention center, as these youth will be assigned a MDFT therapist who will address their mental health and substance abuse issues needs.

Experimental Treatment: Multidimensional Family Therapy-Cross Systems (MDFT-CS). In Stage 1 (in detention) MDFT-CS, the experimental treatment, consists of two major components: standard initial/engagement work with parents in the home and with adolescents in detention (both conducted weekly for the duration of the adolescents stay in detention), plus a state-of-the-art HIV education prevention module based on CDC-endorsed strategies. The in-detention MDFT will be delivered by therapists employed by the University of Miami/ Center for Treatment Research on Adolescent Drug Abuse (CTRADA) who will continue to treat the youth and family after release from detention. In Stage 2, the experimental treatment includes the standard MDFT components (4 overall change units/targets: adolescent, parent, family interaction, and functioning of the family members vis a vis relevant extrafamilial social systems such as school and juvenile justice).

Enhanced Services as Usual (ESAU). In Stage 1 (in detention), ESAU includes two major components - standard drug treatment services that are delivered by detention staff, and state-of-the-art HIV education prevention intervention delivered to all participating youth.

In Stage 2, community drug treatment providers deliver high quality drug treatment on an outpatient basis. To minimize heterogeneity within the comparison condition, and in order to provide better service and treatment tracking opportunities, the study will only use one community based treatment agency to deliver ESAU per locale at each Research Center.

All measures selected are psychometrically strong, sensitive to change, and have been used widely in adolescent substance abuse treatment studies.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 13 and 17
* Be incarcerated in a juvenile detention facility at intake
* Endorse substance abuse problems on the MAYSI or other intake forms
* Have at least one parent figure willing/able to participate in the intervention and research assessments
* Provide informed consent to participate in the study

Exclusion Criteria:

* Mental retardation or pervasive developmental disorders
* Psychotic features
* Current suicidality defined as Ideation + Plan + High intention to carry out plan
* High risk to receive long-term residential placement directly from detention

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2006-04; Primary Completion 2008-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Substance use | Release from detention through the 42-month follow-up
  Timeline Follow-Back Method of Drug and Alcohol Use, Urine analyses for Drug Use, Personal Experiences Inventory and the Adolescent Diagnostic Interview-Light will be used to measure substance use.

SECONDARY OUTCOMES:
Delinquency | Release from detention through the 42-month follow-up
  National Youth Survey Self-Report Delinquency Scale and the Juvenile/Criminal Justice records will be used to measure delinquency
Sexual Risk Behaviors | Release from detention through the 42-month follow-up
  Timeline Followback of Sexual Risk Behaviors, Urine Analyses for Sexually Transmitted Diseases (STDs) and HIV Testing.

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Liddle, EdD, Principal Investigator — University of Miami
Locations (5):
- United States (5):
  - Pinellas Juvenile Detention Center, Clearwater, Florida
  - Operation PAR Inc., Largo, Florida
  - Here's Help, Inc., Miami, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Miami-Dade Juvenile Detention Center, Miami, Florida

REFERENCES:
- [Background] Liddle HA, Dakof GA, Henderson C, Rowe C. Implementation outcomes of Multidimensional Family Therapy-Detention to Community: a reintegration program for drug-using juvenile detainees. Int J Offender Ther Comp Criminol. 2011 Jun;55(4):587-604. doi: 10.1177/0306624X10366960. Epub 2010 Apr 28. PMID 20427547
- [Background] Marvel F, Rowe CL, Colon-Perez L, DiClemente RJ, Liddle HA. Multidimensional family therapy HIV/STD risk-reduction intervention: an integrative family-based model for drug-involved juvenile offenders. Fam Process. 2009 Mar;48(1):69-84. doi: 10.1111/j.1545-5300.2009.01268.x. PMID 19378646
- [Background] Rowe CL, Wang W, Greenbaum P, Liddle HA. Predicting HIV/STD risk level and substance use disorders among incarcerated adolescents. J Psychoactive Drugs. 2008 Dec;40(4):503-12. doi: 10.1080/02791072.2008.10400656. PMID 19283954
- [Derived] Rowe CL, Alberga L, Dakof GA, Henderson CE, Ungaro R, Liddle HA. Family-Based HIV and Sexually Transmitted Infection Risk Reduction for Drug-Involved Young Offenders: 42-Month Outcomes. Fam Process. 2016 Jun;55(2):305-20. doi: 10.1111/famp.12206. Epub 2016 Feb 16. PMID 26879671